CLINICAL TRIAL: NCT03193476
Title: An International, Multicentre, Prospective, Non-interventional Observational Registry for Patients With X-Linked Hypophosphatemia (XLH)
Brief Title: Registry for Patients With X-Linked Hypophosphatemia
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: XLH Registry Version 3.0
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: X-Linked Hypophosphatemia
Keywords: Crysvita; Burosumab; X-linked Hypophosphatemia (XLH); PHEX Gene Mutation; XLH Registry
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an international, multicentre, prospective, non-interventional, observational Registry of patients with X-Linked hypophosphatemia (XLH). The main objective of this XLH Registry is to collect data to characterise the treatment, progression and long-term outcomes of XLH in both adult and paediatric settings.

DETAILED DESCRIPTION:
Methodology

This is an international, multicentre, prospective, non-interventional, observational Registry of patients with X-Linked hypophosphatemia (XLH). The objectives of this XLH Registry is to collect natural history data of XLH to characterise the treatment, progression and long-term outcomes of XLH in both adult and paediatric patients.

This XLH Registry will invite & include patients with XLH, of all ages & gender, irrespective of whether they are on, or not on, a treatment regimen for their XLH.

However, patients who are concurrently participating in an interventional clinical trial, including Investigator-Initiated Studies, are excluded from the XLH Registry, as per the Exclusion Criteria as set in the Protocol. These patients participating in an interventional clinical trial, when their involvement in the trial has ended, will be approached and invited to be included in the XLH Registry.

A subset of the XLH Registry data will be used to fulfil a Post-Authorisation Safety Study (PASS) as requested by the European Medicines Agency's (EMA's) Committee for Medical Products for Human Use (CHMP). Study centres which agree to participate in the PASS will be asked to solicit adverse events on enrolled patients. Not all centres are expected to participate in the PASS. Furthermore, as part of burosumab's Risk Management Plan (RMP), the majority of the safety concerns are being investigated in a Category 3 Post-Authorisation Safety Study (PASS), which uses the XLH Registry. The data source to conduct the PASS is the data collected in the XLH Registry.

All eligible patients at the participating clinics will be asked to participate in the XLH Registry:

* Informed consent will be obtained from adult patients.
* Parental informed consent for the inclusion of a child will be obtained from the child's legally designated representative in line with national guidance.
* Assent will also be sought from children of applicable age in line with national guidance. In all cases the health professional responsible for enrolling the patient into the XLH Registry will assess the appropriateness of gaining assent from an individual at their discretion.

After the patient or legally designated representative has signed the informed consent, the patient data will be recorded in the XLH Registry, including baseline, retrospective and prospective data. Data will be collected using a web-based Electronic Data Capture (EDC) system. A patient identification number will be automatically generated by the system upon enrolment.

No pre-determined follow-up requirements will apply. However, physicians will be prompted to update patient data in the XLH Registry in relation to the patients' visits to the physician. Physicians will be reminded to update the XLH Registry at 12 months after the previous visit information was entered for a patient.

For those patients who attend clinic at more frequent intervals as part of their standard care, data for these visits will be entered at the 12-month intervals with an option to add multiple dates.

This is a prospective observational Registry and no additional interventions other than standard clinical practice are required by the protocol.

ELIGIBILITY:
A patient must meet the following criteria at the enrolment visit (baseline) to be eligible for inclusion into this XLH Registry

Inclusion Criteria:

1. Patients aged from ≥0 years of age at baseline
2. In the opinion of the treating physician the patient has a clinical presentation, radiological, biochemical or genetic investigation results that support diagnosis of XLH
3. Patient is not currently participating in an interventional clinical trial

A patient who meets any of the following criteria at the enrolment visit (baseline) will be excluded from this XLH Registry

Exclusion Criteria:

1. Patient or their legally designated representative does not have the cognitive capacity to provide informed consent.
2. Patient is currently participating in an interventional clinical trial. Patients will be approached for inclusion into the registry once their involvement in the trial ends (including the completion of all trial follow up assessments).
3. Participation in a Compassionate Use Program, Pre-commercial Program (i.e. Named Patient Sales, Nominative ATU) or Investigator Initiated Study does not preclude a patient from participation in this XLH Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with XLH independent of treatment regimen
Sampling Method: Non-Probability Sample
Enrollment: 1343 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 10 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (115):
- Belgium (7):
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
- Bulgaria (2):
  - SHATPD "Prof Ivan Mitev" EAD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
- Czechia (2):
  - Children Hospital, Brno
  - Fakultni nemocnice v Motole, Prague
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Århus Universitetshospital - Aarhus sygehus, Aarhus
  - Århus Universitetshospital, Aarhus
  - Hospital South West Jutland, Esbjerg
  - Rigshospitalet - Paediatric, København Ø
  - Rigshospitalet, København Ø
  - OUH, Odense
- France (11):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux
  - CHU de Lyon - Hôpital Femme Mere Enfant, Bron
  - CHRU Lille, Lille
  - Hopital Roger Salengro - CHU Lille, Lille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital Cochin, Paris
  - CHU Paris Sud - Hopital Bicêtre, Paris
  - Hôpital Bicêtre, Paris
  - "Hopital Pierre-Paul Riquet Centre de Rhumatologie", Toulouse
  - Hopital Purpan, Toulouse
- Germany (8):
  - Klinikum Ernst-von-Bergmann Potsdam und Bad Belzig, Bad Belzig
  - Uniklinikum Bochum, Bochum
  - Uniklinikum Koeln, Cologne
  - MVZ Dr. Eberhard & Partner, Dortmund
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum, Leipzig
  - Hormon and Stoffwechselzentrum, Mainz
- Semmelweis Egyetem, Budapest, Hungary
- The Children's University Hospital, Dublin, Ireland
- Israel (4):
  - Rambam Health Care Center, Haifa
  - Schneider Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Dana-Dwek Children's Hospital, Tel Aviv
- Italy (18):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - AO S. Pio G. Rumno, Benevento
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Presidio Ospedaliero Di Summa Antonio Perrino, Brindisi
  - Azienda Ospedaliera Brotzu, Cagliari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS, Genova
  - ICOT-Istituto Chirurgico Ortopedico Traumatologico, Latina
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Ospedale San Raffaele - Adult, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Istituto Auxologico Italiano -I.R.C.C.S., Piancavallo
  - Stabilimento Ospedaliero Santa Chiara, Pisa
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino (Presidio Sant'Anna), Torino
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - I.R.C.C.S. Burlo Garofolo, Trieste
- Children's Clinical University Hospital, Riga, Latvia
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Norway (3):
  - Oslo University Hospital, Oslo
  - Oslo Universitetssykehus HF, Ulleval, Oslo
  - St. Olav's University Hospital, Trondheim
- Portugal (5):
  - Hospital Pediatrico de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital Dona Estefânia, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo António, Porto
  - Hospital de Sao Joao, Porto
- National Institute of Childrenś Health NUDCH, Bratislava, Slovakia
- University Clinical Centre Ljubljana, Ljubljana, Slovenia
- Spain (11):
  - Hospital de Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Santa Lucía, Cartagena
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
- Sweden (4):
  - Queen Silvia Children's Hospital, Gothenburg
  - Lund University, Lund
  - Karolinska Institute, Stockholm
  - Karolinska Institute (Pediatric), Stockholm
- Switzerland (5):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve (HUG), Geneva
  - Centre Hopitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Klinik Hirslanden Zuerich, Zurich
- United Kingdom (22):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol and Weston, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Royal Hospital for Sick Children and Young People, Edinburgh
  - Gartnavel General Hospital, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Raigmore Hospital, Inverness
  - Leeds General Infirmary, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - National Hospital for Neurology and Neurosurgery, London
  - Evelina Childrens Hospital, London
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Oxford University Hospital NHS Trust, Oxford
  - Sheffield Childrens Hospital, Sheffield
  - Sheffield Teaching Hospitals, Sheffield
  - Southampton General Hospital, Southampton
  - Stanmore Royal Orthopaedic Hospital, Stanmore

REFERENCES:
- [Derived] Carpenter TO, Fukumoto S, Haffner D, Imel EA, Ozono K, Ishii H, Li Z, Sandilands K, Joos-Vandewalle P, Lee C, Kanematsu M, McCullough KP, Brandi ML. Advancing Patient Evidence in XLH (APEX): Baseline analysis of a global data unification program. Bone. 2025 Dec;201:117649. doi: 10.1016/j.bone.2025.117649. Epub 2025 Sep 15. PMID 40962182
- [Derived] Brandi ML, Ariceta G, Beck-Nielsen SS, Boot AM, Briot K, de Lucas Collantes C, Emma F, Giannini S, Haffner D, Keen R, Levtchenko E, Mӓkitie O, Nilsson O, Schnabel D, Tripto-Shkolnik L, Zillikens MC, Liu J, Tudor A, Mughal MZ. Post-authorisation safety study of burosumab use in paediatric, adolescent and adult patients with X-linked hypophosphataemia: rationale and description. Ther Adv Chronic Dis. 2022 Sep 5;13:20406223221117471. doi: 10.1177/20406223221117471. eCollection 2022. PMID 36082134